CLINICAL TRIAL: NCT03053388
Title: Evaluation of the Efficacy Safety and Tolerability of Nitric Oxide Given Intermittently Via Inhalation to Subjects With Bronchiolitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Beyond Air Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AIT_CP_BRONC02.01
Record Dates: First submitted 2017-02-12; First posted 2017-02-15 (Actual); Last update posted 2019-07-09 (Actual); Status verified 2017-02

CONDITIONS: Bronchiolitis
MeSH Terms: conditions — Bronchiolitis | interventions — Nitric Oxide; Palliative Care

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 - Nitric Oxide treatment (Experimental): • Group 1 (NO treatment) - will receive inhalations of 160 ppm NO combined with O2/air for 30 minutes, every 3-4.5 hours, five times a day (24 hours), for up to 5 days (maximum 25 inhalations), in addition to standard supportive treatment.
  Interventions: Drug: Nitric Oxide; Other: Supportive treatment
- Group 2 - Control treatment (Active Comparator): • Group 2 (Control) - will receive inhalations O2/air using the same treatment schedule and equipment as group 1, in addition to standard supportive treatment.
  Interventions: Other: Supportive treatment

INTERVENTIONS:
Drug: Nitric Oxide — Nitric Oxide given via inhalation in cycles
  Arms: Group 1 - Nitric Oxide treatment
Other: Supportive treatment — Supportive treatment (including oxygen)

SUMMARY:
Double blind, randomized multi-center, evaluation of the efficacy, safety and tolerability of Nitric Oxide (NO) given intermittently via inhalation to subjects with acute bronchiolitis.

Bronchiolitis is defined as an infection of the small airways. It is also the most common manifestation of acute lower respiratory infection (ALRI) in early infancy, and is the leading cause of global child mortality.

Nitric Oxide (NO) has been shown to play a critical role in various biological functions, including in the vasodilatation of smooth muscle, neurotransmission, regulation of wound healing and during immune responses to infection with a microbicidal action directed toward various organisms. In the airways, NO is considered to play a key role in the innate immune system in which the first-line of host defense against microbes is built.

The beneficial effect of NO has been shown in different diseases with several options of doses and regimens; newborn with primary pulmonary hypertension showed improvement in oxygenation after 30 minutes of NO treatment at 10-20 ppm, while subjects with adult respiratory distress syndrome demonstrated clinical improvement during NO treatment at 18 and 36 ppm.

In vitro studies suggested that NO, in part per million (ppm) concentrations, possesses antimicrobial and anti-viral activity against a wide variety of phyla including bacteria, viruses, helminthes and parasites.

Safety and tolerability of 160 ppm NO given intermittently via inhalation were shown in a phase II study performed on 2-12 month infants hospitalized with bronchiolitis. According to data no difference in the proportion of adverse events and serious adverse events were detected between subjects treated with NO and subjects treated with standard supportive treatment.

In this study the investigators wish to assess the efficacy of 160 ppm NO given intermittently via inhalation to 0-12 months-old infants hospitalized due to acute bronchiolitis.

Primary objective: Asses the difference in hospital Length of Stay (LOS) between subjects treated with 160 ppm NO combined with standard supportive treatment and subjects treated with standard supportive treatment.

Secondary objectives: Asses the difference in the time required to achieve clinical improvement, a clinical score ≤5 (Modified Tal score) between subjects treated with 160 ppm NO combined with standard supportive treatment and subjects treated with standard supportive treatment. Assess the difference in the time required to achieve sustained 92% oxygen saturation in room air between subjects treated with 160 ppm NO combined with standard supportive treatment and subjects treated with standard supportive treatment. Characterize the safety and tolerability of 160 ppm NO intermittent inhalation treatment as measure by the rate of adverse events.

In this prospective double-blind, randomized multi-Center study the investigators will enroll up to 120 (no less than 80) subjects aged 0-12 months-old, diagnosed with acute bronchiolitis and requiring in-patient hospitalization.

Enrolled subjects will be randomized into 2 groups. Group 1 -Treatment group - Will receive 160 ppm NO given intermittent via inhalation in addition to standard treatment for up to 5 days. Group 2 - will receive ongoing inhalation of the standard treatment for up to 5 days. Between study and after completing all study inhalations the subject will continue to receive the standard treatment. Oxygen (O2), NO, nitrogen dioxide (NO2) and fraction of inspired oxygen (FiO2) delivered to the patient will be continuously monitored.

Treatment administration: Treatment blindness will be kept by separating between un-blinded team members (giving the actual treatment) and blinded team members, and by hiding the NO container and all study related equipment behind a curtain.

All subjects will return for follow-up visits on day 14(+5), 21(+5) days and will be contacted on day 30 (+5) from day of admission to the department.

ELIGIBILITY:
Inclusion Criteria:

1. 1. Pediatric subjects 0-12-months old.

   a. Including subjects born at ≥28 weeks of gestation.
2. Subjects with acute bronchiolitis requiring in-patient hospitalization expected for 24 hours and more.
3. Clinical score of between 7 to 10 at Screening (without oxygen supplementation).
4. Parent/guardian who is willing and able to sign, an informed consent on behalf of the subject.

Exclusion Criteria:

1. 1. Subjects diagnosed with alveolar pneumonia on Chest X-ray (including WBC≥ 15,000/ul, and Temp >39°C).
2. Previous diagnosis of asthma or requirement for asthma medications.
3. Subjects with >2 previous wheezing episodes.
4. History of life-threatening respiratory distress that requires admission to an intensive care unit for treatment.
5. Subjects with history of methemoglobinemia and/or methemoglobin >5% for any cause.
6. Use of an investigational drug within 30 days before enrolment and/or expected to participate in a new study within 90 days.
7. History of frequent epistaxis (>1 episode/month) or significant hemoptysis within 30 days prior to enrolment (≥5 mL of blood in one coughing episode or >30 mL of blood in a 24-hour period.
8. Taken medications such as chronic systemic corticosteroids, CNS stimulants, theophylline or aminophylline, anti-arrhythmic within a certain time period prior to the study.
9. Unable to comply with the study procedures.
10. Underlying genetic disorders (including Cystic fibrosis) or hypotonia.
11. Having the following signs or symptoms: 1) known pulmonary (lung) and/or cardiac (heart) congenital malformations 2) an underlying renal, or liver insufficiency, immunodeficiency, encephalopathy; 3) known or suspected foreign body aspiration.
12. Any reason that, in the opinion of the investigator, may make the subject unfit for this clinical trial.

Max Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 69 (Actual)
Dates: Start 2017-03-05 (Actual); Primary Completion 2018-04-28 (Actual); Study Completion 2018-04-28 (Actual)

PRIMARY OUTCOMES:
Hospital Length of Stay (LOS) | 12 days
  LOS is measured in hours from the time of first treatment dose to the time of physician decision to discharge.

SECONDARY OUTCOMES:
Clinical score of ≤5 (Modified Tal score). | 12 days
  The time in hours from first treatment dose, required to achieve a clinical score of ≤5.
Oxygen saturation (SaO2) ≥92% in room air (without oxygen supplementation) sustained for at least 2 hours | 12 days
  The time in hours from first treatment dose, required to achieve SaO2 ≥92% in room air sustained for at least 2 hours.
Adverse events and NO-related adverse events including methemoglobinemia and nitrogen dioxide levels. | 5 days

CONTACTS AND LOCATIONS:
Locations (10):
- Israel (10):
  - Haemek Medical Center, Afula
  - Barzili Medical Center, Ashkelon
  - Soroka Medical Center, Beersheba
  - Carmel Medical Center, Haifa
  - Rambam Medical Center, Haifa
  - Hadassah Medical Center, Jerusalem
  - Schneider Children's Hospital, Petah Tikva
  - Sheba Medical Center, Ramat Gan
  - Kaplan Medical Center, Rehovot
  - Tel-Aviv Sourasky Medical Center, Tel Aviv

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Goldbart A, Golan-Tripto I, Pillar G, Livnat-Levanon G, Efrati O, Spiegel R, Lubetzky R, Lavie M, Carmon L, Ghaffari A, Nahum A. Inhaled nitric oxide therapy in acute bronchiolitis: A multicenter randomized clinical trial. Sci Rep. 2020 Jun 15;10(1):9605. doi: 10.1038/s41598-020-66433-8. PMID 32541773